CLINICAL TRIAL: NCT06163131
Title: The Effect of Treatment of Emphysema With Endobronchial Valves on the Diaphragm Mobility
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Kirstine Hermann, Principal Investigator, Aarhus University Hospital
Other Study IDs: KH02
Record Dates: First submitted 2023-11-21; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema or COPD
Keywords: Ultrasound; Diaphragm; Endobronchial valves; Endobronchial Lung Volume Reduction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: COPD patients treated with endobronchial valves.

SUMMARY:
In some patients with chronic obstructive pulmonary disease (COPD) the breathlessness is caused by hyperinflation of the lungs. This causes difficulty breathing air out and makes it harder to breath in new air and limits the movement of the diaphram. The diaphragm is the muscle used for breathing between the chest and the stomach. Some of these patients can receive treatment with endobronchial valves, where one-ways are inserted into the bronchial system the let out some of the excess air, and thereby relieve breathlessness.

The goal of this observational study is to investigate the effect of endobronchial valves on the mobility of the diaphragm in patients with chronic obstructive pulmonary disease. The main questions it aims to answer are:

* If the movement of the diaphragm improves after treatment with endobronchial valves.
* If there is a link between improvement of diaphragm function and improvement of symptoms, lung function and physical ability.
* If ultrasound scan immediately after the treatment will predict which patients will benefit from the treatment.

Participants will undergo ultrasound before, 1 day after and 90 days after the procedure, and lung function examinations from their already planned control visits will be collected.

DETAILED DESCRIPTION:
When emphysema is present in COPD-patients, the impaired expiratory ventilation causes lung hyperinflation. This results in a change in the respiratory mechanisms of the thorax and thereby impairment of the movement capacity of the muscles. The most important respiratory muscle, the diaphragm, is caudally displaced and flattened, hence, the capacity and mobility of the muscle decreases.

Some patients with COPD fulfill the criteria for treatment with endobronchial valves (EBV) where one-way valves can be inserted in the bronchial system. The mechanism behind the effect of EBV is believed to be formation of an atelectasis of the designated lobe and thereby reduction of hyperinflation and hence reduction of symptoms and increase in pulmonary function

In this study the aim is to assess:

1. If the movement of the diaphragm improves after insertion of endobronchial valves in patients with severe emphysema.
2. If there is a correlation between improvement of diaphragm function and improvement of symptoms, lung function examinations and physical ability after insertion of endobronchial valves.
3. If immediate post-procedural ultrasound evaluation of diaphragm function predicts the development of atelectasis and hence clinical outcome

ELIGIBILITY:
Inclusion Criteria:

1. Patients selected to receive treatment with endobronchial valves
2. Signed informed consent

Exclusion Criteria:

1. Neuromuscular disease interfering with diaphragm function
2. Pleural effusion at time of preoperative or 90-days postoperative ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD approved for treatment with endobronchial valves. The suitability will be assessed during multidiciplinary team conference, independent of this study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-11-27 (Estimated); Primary Completion 2026-11-27 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Diaphragm mobility | Before the procedure, 1 day after the procedure and 90 days after the procedure
  The area method[13] will be used for assessment of diaphragm movement, using a curvilinear probe (2-6 MHz). Measurements will be performed during tidal respiration, deep respiration, sniff excursion and constant flow with constant volume, using test flute with bag of air attached.
Diaphragm mobility | Before the procedure, 1 day after the procedure and 90 days after the procedure
  M-mode: Diaphragm excursion in tidal, deep and sniff inspiration will be evaluated in the right side using M-mode through anterior subcostal midclavicular view. Contraction and relaxation velocity will be measured.
Diaphragm Thickening | Before the procedure, 1 day after the procedure and 90 days after the procedure
  Thickness and thickening ratio: The thickness and thickening ratio will be evaluated in B-mode using the linear probe, though lateral intercostal view during tidal respiration.

SECONDARY OUTCOMES:
Forced expiratory volume in 1 second in litres | Before and 90 days after the procedure
  Patients will undergo lung function examinations as a part of the independent preoperative and postoperative assessments
Forced expiratory volume in 1 second % of expected | Before and 90 days after the procedure
  Patients will undergo lung function examinations as a part of the independent preoperative and postoperative assessments
Forced vital capacity in litres | Before and 90 days after the procedure
  Patients will undergo lung function examinations as a part of the independent preoperative and postoperative assessments
Forced vital capacity in % of expected | Before and 90 days after the procedure
  Patients will undergo lung function examinations as a part of the independent preoperative and postoperative assessments
Total lung volume in % of expected | Before and 90 days after the procedure
  Patients will undergo lung function examinations as a part of the independent preoperative and postoperative assessments
Residual volume in % of expected | Before and 90 days after the procedure
  Patients will undergo lung function examinations as a part of the independent preoperative and postoperative assessments
diffusion capacity in % of expected | Before and 90 days after the procedure
  Patients will undergo lung function examinations as a part of the independent preoperative and postoperative assessments
6 Minute walking test | Before and 90 days after the procedure
  Patients will undergo 6 minutes walking test as a part of the independent preoperative and postoperative assessments
Rate of atelectasis on Lung X-ray | Before, one day and 90 days after the procedure
  Patients will receive x ray of the lungs as a part of the independent preoperative and postoperative assessments
Medical Research Council (MRC) Dyspnoea Scale | Before, one day and 90 days after the procedure
  Medical Research Council (MRC) score will be used for symptom burden assessment
COPD Assessment Test (CAT) Score | Before, one day and 90 days after the procedure
  CAT score will be used for symptom burden assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided